CLINICAL TRIAL: NCT00000209
Title: Buprenorphine Dosing Interval
Brief Title: Buprenorphine Dosing Interval - 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-06082-5; R18-06082-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 1994-09

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to explore the feasibility of extending the dosing interval of well maintained buprenorphine patients to 48 and 72 hours, leading to eventual 3 times/week dosing.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Opiate dependence according to DSM-IV critera. Self-reported use within the last 30 days. Agreeable to conditions of study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative-hynotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1992-11

PRIMARY OUTCOMES:
Drug use
Withdrawal symptoms
Opiate and cocaine craving

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States

REFERENCES:
- [Background] 1) Buprenorphine as a pharmacotherapy for opiate addiction. What dose provides a therapeutic response? (An J Add 1996; 5(3): 220-222). (1) Buprenorphine as a pharmacotherapy for opiate addiction. What dose provides a therapeutic response? (An J Add 1996; 5(3):220-222).